CLINICAL TRIAL: NCT06845475
Title: Effect of Shock Wave Therapy on Myofascial Pain Syndrome in Adolescent Athletes
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Hafez Mohamed, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005356
Record Dates: First submitted 2025-02-20; First posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Myofascial Pain Syndrome
MeSH Terms: conditions — Myofascial Pain Syndromes | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Designed physical therapy program (Active Comparator): It will consist of 20 adolescents, who will receive a designed physical therapy program for the treatment of Myofascial pain syndrome.
  Interventions: Other: Designed physical therapy program
- Designed physical therapy program + Extracorporeal shock wave therapy (ESWT) (Experimental): It will consist of 20 adolescents, who will receive the same designed physical therapy program in addition to extracorporeal shock wave therapy (ESWT).
  Interventions: Other: Designed physical therapy program; Other: Extracorporeal shock wave therapy (ESWT)

INTERVENTIONS:
Other: Designed physical therapy program — Both groups will receive a designed physical therapy program, in the form of myofascial trigger points pressure release, stretching of the upper trapezius muscle, strengthening exercises, and infrared radiation for 4 weeks.
Other: Extracorporeal shock wave therapy (ESWT) — Adolescents of the experimental group will receive Extracorporeal shock wave therapy with the following parameters; low-level energy radial extracorporeal shock wave by (STORZ MEDICAL Master Pulse MP200), each subject received 3 sessions per week for 4 weeks with 700 impulse/session 400 impulse was applied to tight band and 300 impulses will be applied surrounding the tight band, with frequency [10HZ], resulting in positive energy flux density [EFD] 0.056mJ/mm.
  Arms: Designed physical therapy program + Extracorporeal shock wave therapy (ESWT)

SUMMARY:
The purpose of the study is to determine the effect of extracorporeal shockwave therapy on pain, neck range of motion, and functional activity in adolescent athletes.

DETAILED DESCRIPTION:
Myofascial pain syndrome is a syndrome characterized by pain and accompanying muscle spasms, referred pain patterns, stiffness, and restricted range of motion caused by trigger points on constricted fibers of muscles and/or fasciae. Myofascial pain syndrome is the most common reason for back pain, shoulder pain, tension-type headaches, and regional pains such as facial pain.

Myofascial trigger points (MTrPs) are understood as the morphological correlate of the myofascial pain syndrome (MPS), an acute or chronic muscular pain condition affecting a single muscle or a group of muscles. Active MTrPs are spontaneously painful, while latent MTrPs are only painful upon pressure. MTrP stimulation can also cause referred pain and the characteristic local twitch response.

The main goal of MPS treatment is to break down the vicious circle of "spasm - pain - spasm" and release trigger points. Various physical therapy modalities such as trigger point injection, stretching-spray technique or ultrasound (US), heat packs and transcutaneous electrical nerve stimulation (TENS), and extracorporeal shock wave therapy (ESWT), are used for the treatment of MPS. These modalities inactivate the trigger point with their thermal and mechanical effects.

Due to the lack of research area of extracorporeal shock wave therapy on myofascial pain syndrome on upper trapezius in adolescents' athletes, so the purpose of the study is to know impact of the extracorporeal shock wave therapy on myofascial pain syndrome on upper trapezius in adolescents' athletes.

ELIGIBILITY:
Inclusion Criteria:

* Age ranges from 14 to 18 years.
* All adolescents have regional pain complaint.
* Tenderness in cervical trigger points in the midpoint of the upper border of the trapezius muscle, from grade 2 to grade 4 according to the tenderness grading scheme (Hubbard, 1993) (Appendix II).
* Palpation of a trigger point elicits a stereotypic zone of referred pain specific to that muscle.
* Identification of a palpable taut band, as well as a palpable, and exquisitely tender spot along the length of that taut band.
* All adolescents are allowed to practice their regular sports activities.

Exclusion Criteria:

* Dermatological disorders.
* Having myofascial trigger points injection.
* Chronic pain in both sides of the body.
* History of findings of cervical injury whether orthopedic or soft tissue injury.
* Analgesic drugs or NSAIDs during the treatment period.

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-02-25 (Estimated); Primary Completion 2025-04-25 (Estimated); Study Completion 2025-05-05 (Estimated)

PRIMARY OUTCOMES:
Assessment of pain level | 4 weeks
  By Pain Quality Assessment Scale (PQAS), which help to measure different aspects of pain. For one patient, a pain might feel extremely hot and burning, but not at all dull, while another patient may not experience any burning pain, but feel like their pain is very dull and achy. High test-retest reliability has been observed in both literate and illiterate patients with neuropathic pain, for construct validity, was high in patients with chronic pain conditions. The scale creates a 20- item measures that would be even more useful for assessing neuropathic pain and also would be used to assess pain qualities associated with non-neuropathic pain. PQAS can be scored as individual ratings (20 items), or the PQAS items can be combined into composite scores.

SECONDARY OUTCOMES:
Assessment cervical flexion range of motion (ROM) | 4 weeks
  It will be assessed by the CROM instrument pre and post-treatment. The subject should be seated upright in a straight-back chair with the sacrum against the backrest, thoracic spine away, arms at the sides, and feet flat on the floor. The CROM instrument is positioned like a pair of glasses and secured with Velcro straps. To ensure full cervical flexion, the movement begins with a slight nod to create a double chin (suboccipital flexion) before continuing into full flexion. The sagittal plane meter should be read through its beveled edge for an accurate magnified reading, and the measurement is recorded on the designated sheet.
Assessment cervical extension range of motion (ROM) | 4 weeks
  It will be assessed by the CROM instrument pre and post-treatment. Cervical extension is measured by initiating a slight backward nod (suboccipital extension), followed by further extension until the full range is reached. The obtained measurement is then recorded accordingly.
Assessment cervical lateral flexion ROM to the right | 4 weeks
  It will be assessed by the CROM instrument pre and post-treatment. To prevent rotation during lateral flexion, focus should remain on a fixed point straight ahead. A sagittal plane meter reading of zero confirms a neutral head position, while any deviation on the lateral flexion meter indicates lateral flexion at rest, which should be recorded. Lateral flexion of the head to the right is performed while maintaining level shoulders and avoiding rotation. Shoulder elevation is monitored and corrected manually if needed.
Assessment cervical lateral flexion ROM to the left | 4 weeks
  It will be assessed by the CROM instrument pre and post-treatment. To prevent rotation during lateral flexion, focus should remain on a fixed point straight ahead. A sagittal plane meter reading of zero confirms a neutral head position, while any deviation on the lateral flexion meter indicates lateral flexion at rest, which should be recorded. Lateral flexion of the head to the left is performed while maintaining level shoulders and avoiding rotation. Shoulder elevation is monitored and corrected manually if needed.
Assessment cervical rotation ROM to the right | 4 weeks
  It will be assessed by the CROM instrument plus the magnetic yoke and rotation arm pre and post-treatment. Accurate readings depend on determining magnetic north by observing the red needle on the rotation meter at least four feet from the yoke. The magnetic yoke is positioned on the subject's shoulders with the arrow pointing north. The subject remains seated upright in a straight-back chair with the sacrum against the backrest, thoracic spine away, arms at the sides, and feet flat. The lateral flexion and sagittal plane meters must read zero to ensure a level rotation meter. With the subject facing forward, the rotation meter is adjusted so one pointer aligns with zero. A fixed horizontal line on the wall serves as a visual reference to prevent head tilting. Rotation to the right occurs first, with the left shoulder lightly stabilized to prevent movement.
Assessment cervical rotation ROM to the left | 4 weeks
  It will be assessed by the CROM instrument plus the magnetic yoke and rotation arm pre and post-treatment. Accurate readings depend on determining magnetic north by observing the red needle on the rotation meter at least four feet from the yoke. The magnetic yoke is positioned on the subject's shoulders with the arrow pointing north. The subject remains seated upright in a straight-back chair with the sacrum against the backrest, thoracic spine away, arms at the sides, and feet flat. The lateral flexion and sagittal plane meters must read zero to ensure a level rotation meter. With the subject facing forward, the rotation meter is adjusted so one pointer aligns with zero. A fixed horizontal line on the wall serves as a visual reference to prevent head tilting. Rotation to the left occurs first, with the right shoulder lightly stabilized to prevent movement.
Assessment of functional activity of neck | 4 weeks
  It will be assessed pre and post-treatment using the neck disability index (NDI).The 10 items include effects of pain on personal care activities: lifting, reading, sleeping and the patient level of participation in recreational activities. Each section contains 6 statements representing a different level of severity. Each section is scored on a 0 to 5 scale, with 5 designating the greatest disability. The scores of each section are summated for a total score of 50. The total score is then multiplied by 2 to arrive at percentage score. This value represents the percentage of disability.

CONTACTS AND LOCATIONS:
Overall Officials: Nanees Essam Mohamed Salem, PhD, Study Chair — Professor, Cairo university
Locations (1):
- Ismailia Medical Complex, Ismailia, Egypt